CLINICAL TRIAL: NCT05966142
Title: A Depression and Opioid Pragmatic Trial in Pharmacogenetics
Brief Title: A Depression and Opioid Pragmatic Trial in Pharmacogenetics (Chronic Pain Trial)
Acronym: ADOPT PGx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); University of Florida (Other); Vanderbilt University Medical Center (Other); Indiana University School of Medicine (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00104948_B; U01HG010225 (NIH)
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain
Keywords: Pharmacogenetic; CYP2D6; CYP2C19
MeSH Terms: conditions — Chronic Pain | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: Immediate vs. delayed pharmacogenetic testing and genotype-guided pain or depression therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Pain - Immediate PGx Testing (Experimental): Immediate genetic testing of CYP2D6 and clinical decisions support for pain management prescribing to the healthcare provider
  Interventions: Other: Pharmacogenetic testing; Other: Clinical decisions support
- Chronic Pain - Delayed PGx Testing (Other): Delayed genetic testing of CYP2D6 and return of results after the conclusion of the 6-month follow-up period
  Interventions: Other: Pharmacogenetic testing

INTERVENTIONS:
Other: Pharmacogenetic testing — Genetic testing of CYP2D6 and CYP2C19
Other: Clinical decisions support — Prescribing recommendations to the provider based on the pharmacogenetic testing results
  Arms: Chronic Pain - Immediate PGx Testing

SUMMARY:
This study is comprised of three separate pharmacogenetic trials grouped into a single protocol due to similarities in the intervention, the hypotheses, and the trial design. The three trials are the Acute Pain Trial, the Chronic Pain Trial, and the Depression Trial. Participants can enroll in only one of the three trials. All three trials were registered on ClinicalTrials.gov under NCT04445792. In July 2023 each of the three treatment trials was registered under a separate NCT# and NCT04445792 was converted to a screening record per recent guidance on master protocol research programs (MPRPs). This record is specific to the Chronic Pain Trial within the ADOPT-PGx protocol.

The Chronic Pain Trial is a prospective, multicenter, two arm randomized pragmatic trial. Participants meeting eligibility criteria will be randomly assigned to either immediate pharmacogenetic testing and genotype-guided opioid therapy (Intervention arm) or standard care with 6-month delayed pharmacogenetic testing (Control arm). The investigators will test the hypothesis that pharmacogenetic testing and genotype guided pain therapy improves pain control after surgery in participants who's body processes some pain medicines slower than normal.

DETAILED DESCRIPTION:
Pain and depression are conditions that impact substantial proportions of the US population. Finding safe and effective drug therapies for both conditions is challenging. In the case of treatment for acute and chronic pain, the challenge is finding effective therapy while minimizing adverse effects or opioid addiction (and the ensuing consequences). For depression, there are few clinically relevant predictors of successful treatment leading to multiple trials of inadequate therapy for some patients. Both opioid and antidepressant prescriptions can be guided by pharmacogenetics (PGx) data based on existing guidelines from the Clinical Pharmacogenetics Implementation Consortium (CPIC).

This study is designed to evaluate the impact of pharmacogenetic testing and genotype-guided pain or anti-depressant therapy on pain control or depression symptoms in a pragmatic setting.

The rationale for examining a genotype-guided approach to acute and chronic pain management is based on the importance of CYP2D6 for the bioactivation of tramadol, codeine, and hydrocodone and data from a pilot study supporting improved pain control in intermediate and poor CYP2D6 metabolizers in the genotype-guided arm who are taking these drugs at baseline. Similarly, the rationale for examining a genotype-guided approach to depression medication therapy is based on the demonstrated role of CYP2D6 in the bio inactivation and CYP2C19 oxidation of select, commonly used SSRIs. Secondly, data from industry sponsored trials support the hypothesis of improved depression symptom control in a genotype-guided arm.

Study objectives:

Determine if a genotype-guided approach to pain therapy in participants with at least 3 months of chronic pain leads to improved pain control compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

Chronic Pain Trial

* Age ≥ 18 years
* English speaking or Spanish speaking
* Seen at primary care clinics (such as, but not limited to, Internal Medicine, Family Medicine or Pediatrics) or patients seen in pain-relevant specialty clinics
* History of pain for at least the last 3 months
* Currently treated or being considered for treatment with tramadol, hydrocodone, or codeine to improve pain management

Exclusion Criteria

Trial-wide:

* Life expectancy less than 12 months
* Are too cognitively impaired to provide informed consent and/or complete study protocol
* Are institutionalized or too ill to participate (i.e. mental or nursing home facility or incarcerated)
* Have a history of allogeneic stem cell transplant or liver transplant
* People with prior clinical pharmacogenetic test results for genes relevant for the study in which they will enroll (CYP2D6 for the pain studies and CYP2D6 or CYP2C19 for depression) or already enrolled in an ADOPT PGx trial

Chronic Pain

* Plan to move out of the area within 6 months of enrollment
* Undergoing treatment for an active cancer diagnosis
* Currently taking daily opioids other than tramadol, codeine or hydrocodone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1048 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hrishikesh Chakraborty, Study Director — Duke University; Todd Skaar, PhD, Principal Investigator — Indiana University
Locations (10):
- United States (10):
  - University of Florida - Gainesville, Gainesville, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Institute for Family Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Meharry Medical College, Nashville, Tennessee
  - Nashville General Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skaar TC, Myers RA, Fillingim RB, Callaghan JT, Cicali E, Eadon MT, Elwood EN, Ginsburg GS, Lynch S, Nguyen KA, Obeng AO, Park H, Pratt VM, Rosenman M, Sadeghpour A, Shuman S, Singh R, Tillman EM, Volpi S, Wiisanen K, Winterstein AG, Horowitz CR, Voora D, Orlando L, Chakraborty H, Van Driest S, Peterson JF, Cavallari LA, Johnson JA, Dexter PR; IGNITE Pragmatic Trials Network. Implementing a pragmatic clinical trial to tailor opioids for chronic pain on behalf of the IGNITE ADOPT PGx investigators. Clin Transl Sci. 2024 Aug;17(8):e70005. doi: 10.1111/cts.70005. PMID 39177194
- See also: Implementing a pragmatic clinical trial to tailor opioids for chronic pain on behalf of the IGNITE ADOPT PGx investigators — http://pubmed.ncbi.nlm.nih.gov/39177194/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This record is specific to the Chronic Pain Trial within the ADOPT PGx protocol. It only contains the participants consented to the Chronic Pain Trial.
Pre-assignment Details: There were 1092 participants consented into the Chronic Pain trial. Of the 1092, 44 were not randomized into the trial and were not assigned to a treatment arm. The remaining 1048 consented participants were randomized and assigned into the treatment arms. The 1048 randomized participants will be described moving forward.
Period: Overall Study
Arm/Group | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing
Started | 527 | 521
Completed | 456 | 457
Not Completed | 71 | 64
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 55 | 52
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Duplicate Enrollment | 1 | 0
Not completed — Study Logistical Reason | 1 | 0
Not completed — Unable to complete follow up due to change in health | 1 | 1

BASELINE CHARACTERISTICS:
Population: ITT refers to the Intent To Treat population, while mITT, a subset of ITT, refers to the modified Intent To Treat population. The mITT population is the primary analytical population for the Chronic Pain Trial and includes participants who have a CYP2D6 activity scores <= 0.75 after accounting for CYP2D6 phenoconversion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing | Total
Number analyzed (Participants) | 527 | 521 | 1048
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Intent to Treat (ITT) population
  years | 58.2 (12.2) | 57.8 (11.9) | 58.0 (12.1)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Modified Intent to Treat (mITT) population
  years
    number analyzed (Participants) | 136 | 146 | 282
    (all) | 58.0 (10.9) | 57.8 (11.3) | 57.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Intent to Treat (ITT) population. Three participants declined to answer.
  Participants
    number analyzed (Participants) | 524 | 521 | 1045
    Female | 373 | 375 | 748
    Male | 151 | 146 | 297
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Modified Intent to Treat (mITT) population. Two participants declined to answer.
  Participants
    number analyzed (Participants) | 134 | 146 | 280
    Female | 95 | 115 | 210
    Male | 39 | 31 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Intent to Treat (ITT) population
  Participants
    Hispanic or Latino | 48 | 45 | 93
    Not Hispanic or Latino | 468 | 469 | 937
    Unknown or Not Reported | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Modified Intent to Treat (mITT) population
  Participants
    number analyzed (Participants) | 136 | 146 | 282
    Hispanic or Latino | 13 | 12 | 25
    Not Hispanic or Latino | 119 | 131 | 250
    Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Intent to Treat (ITT) population
  Participants
    American Indian or Alaska Native | 6 | 7 | 13
    Asian | 2 | 7 | 9
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 207 | 201 | 408
    White | 245 | 245 | 490
    More than one race | 13 | 17 | 30
    Unknown or Not Reported | 53 | 44 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Modified Intent to Treat (mITT) population
  Participants
    number analyzed (Participants) | 136 | 146 | 282
    American Indian or Alaska Native | 2 | 1 | 3
    Asian | 2 | 5 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 49 | 48 | 97
    White | 66 | 75 | 141
    More than one race | 2 | 6 | 8
    Unknown or Not Reported | 15 | 11 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 527 | 521 | 1048

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity
Description: The composite pain intensity score is derived from the 3-time PROMIS (Patient-Reported Outcomes Measurement Information System) pain intensity scale. Composite pain intensity score is the sum of the 3 questions and ranges from 3 (no pain) to 15 (intense pain). Change in composite pain intensity score ranges from -12 (change from the highest level of pain to the lowest level of pain) to 12 (change from the lowest level of pain to the highest level of pain).
Time Frame: Baseline to 3 months
Population: Modified Intent to Treat (mITT) population with completed baseline and 3-month pain surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing
Number analyzed (Participants) | 125 | 130
score on a scale | -0.7 (2.3) | -0.8 (2.4)
Statistical Analysis 1: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.5913, t-test, 2 sided; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.42 to 0.74]

2. Secondary Outcome: Pain Reduction Magnitude
Description: Ratio of Composite Pain Score at 3 months relative to baseline. Composite pain intensity scores were shifted to range 0-12 and the pain reduction magnitude is reported as the ratio of pain at 3 months relative to pain at baseline using this adjusted scale. Statistical analyses were conducted using the log ratio pain at 3 months relative to pain at baseline. Due to the presence of 0 values in the ratios, the log ratios include a +.5 offset, i.e. log(3-month pain +.5 / baseline pain + 0.5).
Time Frame: Baseline to 3 months
Population: Modified Intent to Treat (mITT) population with completed baseline and 3-month pain surveys.
Measure: Mean (Standard Deviation); unit: log ratio
Arm/Group | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing
Number analyzed (Participants) | 125 | 130
log ratio | -0.1 (0.4) | -0.1 (0.5)
Statistical Analysis 1: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.6803, t-test, 2 sided

3. Secondary Outcome: Number of Participants With Clinically Significant Pain Reduction
Description: Clinically significant pain reduction defined as ratio of 3-month composite pain score relative to baseline is < 0.7, corresponding to a 30% or more improvement in pain scores.
Time Frame: Baseline to 3 months
Population: Modified Intent to Treat (mITT) population with completed baseline and 3-month pain surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing
Number analyzed (Participants) | 125 | 130
Participants | 17 | 27
Statistical Analysis 1: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.1228, Chi-squared

4. Secondary Outcome: Prescription Pain Medication Misuse as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: The 7-item PROMIS questionnaire assesses the extent to which participant experience prescription pain medication misuse symptoms in the past 3 months using a 5-point Likert scale. Participants are asked if they have had a prescription for pain medication in the last 3 months. If no, the questionnaire is not administered, if yes, the questionnaire is administered. For the completed questionnaires. Raw scores ranging from 7 to 35. Raw scores are converted to T-scores using the PROMIS conversion table, with T-scores ranging 36.3 to 54.1. Higher T-scores reflect greater symptom severity.
Time Frame: 3 months
Population: Modified Intent to Treat (mITT) participants who indicate having taken a prescription for pain medication in the past 3 months.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing
Number analyzed (Participants) | 106 | 109
T-score | 40.1 (4.8) | 40.5 (4.8)
Statistical Analysis 1: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.5252, t-test, 2 sided; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.7 to 0.9]

5. Secondary Outcome: Number of Participants With Drug-Gene Concordance
Description: Concordance between the participant reported opioid medications at 3 months and CYP2D6 phenotype.
Time Frame: 3 months
Population: Modified Intent to Treat (mITT) participants with prescription pain medication data collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing
Number analyzed (Participants) | 123 | 133
Participants | 33 | 36
Statistical Analysis 1: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.9657, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Per the study protocol, only Adverse Device Effect (ADE) events suspected to be related to the specimen collection, laboratory assay genotyping results, and phenoconversion recommendations from the Best Practice Alerts (BPAs)/Consult notes were reported to the IRB. Reportable ADEs or unanticipated Adverse Device Effect (UADEs) events including unanticipated study related deaths will be collected in the study database per IRB reporting policies. Medication side effects were not included as AEs.
Arm/Group | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing
All-Cause Mortality (participants affected / at risk) | 3/527 | 3/521
Serious Adverse Events (participants affected / at risk) | 0/527 | 0/521
Other Adverse Events (participants affected / at risk) | 0/527 | 0/521

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/42/NCT05966142/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT05966142/ICF_000.pdf